CLINICAL TRIAL: NCT00859274
Title: Saline Challenge in Monitoring Asthma Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Heikki Koskela, Respiratory Physician, Kuopio University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KUH5801112
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Budesonide (Experimental): All patients receive this treatment to induce a change in asthma control
  Interventions: Drug: budesonide

INTERVENTIONS:
Drug: budesonide — Budesonide is given via inhalation utilising a dry powder inhaler called Easyhaler. The dosage is 400 ug twice daily. The duration of the study is 12 weeks but very probably the patients continue the usage of this drug as a part of their routine clinical management.

SUMMARY:
It is generally accepted that symptoms and lung function are not sufficient ways to monitor asthma control. Therefore, several objective tests have been developed to help asthma control monitoring, each having their own shortcomings. We have developed a new test, the hypertonic saline cough challenge. In our previous publication this test has proven useful in diagnosing asthma. The present study is planned to investigate whether hypertonic saline cough challenge could be used to monitor asthma control. A group of steroid-naive asthmatics will be recruited. A treatment with inhaled budesonide is started. Asthma control is monitored at regular intervals utilising a validated questionnaire. At the same time points, hypertonic saline cough challenges will be performed. We will analyse whether changes in the responsiveness to the cough challenge reflects the changes in asthma control

ELIGIBILITY:
Inclusion Criteria:

* symptomatic asthma

Exclusion Criteria:

* usage of inhaled or oral corticosteroids
* recent febrile respiratory infection
* severe, unstable asthma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Changes in responsiveness to hypertonic saline cough challenge | Before budesonide treatment, and after 1, 4, and 12 weeks' treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory Medicine, Kuopio University Hospital, Kuopio, Finland

REFERENCES:
- [Derived] Koskela HO, Purokivi MK. Airway oxidative stress in chronic cough. Cough. 2013 Dec 2;9(1):26. doi: 10.1186/1745-9974-9-26. PMID 24294924
- [Derived] Koskela HO, Purokivi MK. Capability of hypertonic saline cough provocation test to predict the response to inhaled corticosteroids in chronic cough: a prospective, open-label study. Cough. 2013 May 20;9:15. doi: 10.1186/1745-9974-9-15. eCollection 2013. PMID 23688169